CLINICAL TRIAL: NCT00428883
Title: Rare Disease With Microvascular Involvement: High Dose Intravenous N-Acetylcysteine Versus Iloprost for Early, Rapidly Progressive Diffuse Systemic Sclerosis
Brief Title: High Dose Intravenous N-Acetylcysteine Versus Iloprost for Early, Rapidly Progressive Diffuse Systemic Sclerosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Politecnica delle Marche (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FARM5X8AWM
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Scleroderma, Diffuse
Keywords: Scleroderma, Systemic; Scleroderma, Diffuse
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine (NAC)

SUMMARY:
* Systemic sclerosis (scleroderma; SSc) is a rare, disfiguring systemic disorder characterized by fibrosis of the skin and visceral organs that alters every aspect of an individual life
* Although some features of scleroderma phenotype are well established and represent the hallmarks of the disease, the primary cause is not fully delineated, though both endothelial cell damage, immunological abnormalities and excessive extracellular matrix production are well-documented
* Recently, excessive oxidative stress has been implicated in the pathogenesis of scleroderma
* N-acetylcysteine (NAC) exhibits direct and indirect antioxidant properties. Its free thiol group is capable of interacting with the electrophilic groups of ROS. This interaction with ROS leads to intermediate formation of NAC thiol, with NAC disulphide as a major end product. The net result is a decrease of the concentrations of OH-, H2O2, and HOCl. In addition, NAC exerts an indirect antioxidant effect related to its role as a glutathione (GSH) precursor. It serves as a central factor in protecting against internal toxic agents.
* In view of these considerations we expect that NAC can confer substantial benefit in patients with scleroderma reducing skin fibrosis in view of its antioxidant properties, and we have decided to conduct a double blind, multicenter trial to establish whether NAC could ameliorate skin fibrosis in scleroderma patients

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of early diffuse scleroderma
* ability to give an informed consent
* use of an acceptable method of birth control (if women in childbearing age). Pregnancy will be ruled out before study beginning.

Exclusion Criteria:

* connective tissue diseases or other autoimmune diseases other than SSc;
* history of intolerance to the study drugs;
* severe cardiac failure (NYHA >=3 or left ventricular ejection fraction <40%), recent (<6 months) history of myocardial infarction; symptomatic ischemic myocardial disease, ventricular tachyarrhythmia, atrial fibrillation;
* resting PaO2 <60mm/hg
* creatinine clearance below 90ml/h
* severe hepatic failure
* bronchial asthma h. hemorrhagic diathesis i. pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2007-01; Study Completion 2009-02

PRIMARY OUTCOMES:
The primary outcome is the reduction of skin thickness
Evaluated by the modified Rodnan skin score.

SECONDARY OUTCOMES:
scleroderma disease activity assessed as established
patient physical and emotional well-being (VAS, HAQ, SF36)
laboratory evidence of skin fibroblast activation;
the levels of Glutathione and of oxidized glutathione (GSSG).

CONTACTS AND LOCATIONS:
Overall Officials: Armando Gabrielli, MD,professor, Principal Investigator — Università Politecnica delle Marche
Locations (5):
- Italy (5):
  - Università politecnica delle marche, Ancona
  - Università di Firenze, Florence
  - Università de L'Aquila, L’Aquila
  - Seconda Università di Napoli, Napoli
  - Catholic University of the Sacred, Roma